CLINICAL TRIAL: NCT04482725
Title: A Trial to Assess the Injection Site Pain Experience of Excipient Solutions Relevant for Subcutaneous Injection
Brief Title: Injection Site Pain Comparison of Excipient Solutions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: NN9838-4703; U1111-1250-7817 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- S1 (Experimental): Day 1: Trial products 1-2-12-3-11-4 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 10-5-9-6-8-7 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S2 (Experimental): Day 1: Trial products 2-3-1-4-12-5 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 11-6-10-7-9-8 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S3 (Experimental): Day 1: Trial products 3-4-2-5-1-6 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 12-7-11-8-10-9 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S4 (Experimental): Day 1: Trial products 4-5-3-6-2-7 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 1-8-12-9-11-10 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S5 (Experimental): Day 1: Trial products 5-6-4-7-3-8 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 2-9-1-10-12-11 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S6 (Experimental): Day 1: Trial products 6-7-5-8-4-9 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 3-10-2-11-1-12 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S7 (Experimental): Day 1: Trial products 7-8-6-9-5-10 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 4-11-3-12-2-1-given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S8 (Experimental): Day 1: Trial products 8-9-7-10-6-11 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 5-12-4-1-3-2 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S9 (Experimental): Day 1: Trial products 9-10-8-11-7-12 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 6-1-5-2-4-3 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S10 (Experimental): Day 1: Trial products 10-11-9-12-8-1 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 7-2-6-3-5-4 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S11 (Experimental): Day 1: Trial products 11-12-10-1-9-2 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 8-3-7-4-6-5 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12
- S12 (Experimental): Day 1: Trial products 12-1-11-2-10-3 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Day 2: Trial products 9-4-8-5-7-6 given as subcutaneous injections (s.c., under the skin) on alternate sides of the abdomen.
  Interventions: Other: Trial product 1; Other: Trial product 2; Other: Trial product 3; Other: Trial product 4; Other: Trial product 5; Other: Trial product 6; Other: Trial product 7; Other: Trial product 8; Other: Trial product 9; Other: Trial product 10; Other: Trial product 12

INTERVENTIONS:
Other: Trial product 1 — Buffering agent: N/A Isotonic agent: NaCl 9.0 mg/mL
Other: Trial product 2 — Buffering agent: Disodium hydrogen phosphate, dihydrate 1.42 mg/mL Isotonic agent: NaCl 8.25 mg/mL
Other: Trial product 3 — Buffering agent: Disodium hydrogen phosphate dihydrate 1.42 mg/mL Isotonic agent: Propylene glycol 18.5 mg/mL
Other: Trial product 4 — Buffering agent: Disodium hydrogen phosphate dihydrate 1.42 mg/mL Isotonic agent: Glycerol 22.0 mg/mL
Other: Trial product 5 — Buffering agent: Disodium hydrogen phosphate dihydrate 1.42 mg/mL Isotonic agent: Mannitol 44.0 mg/mL
Other: Trial product 6 — Buffering agent: Disodium hydrogen phosphate dihydrate 1.42 mg/mL Isotonic agent: Sucrose 82.0 mg/mL
Other: Trial product 7 — Buffering agent: Disodium hydrogen phosphate dihydrate 1.42 mg/mL Isotonic agent: a,a-Trehalose, dihydrate 90.0 mg/mL
Other: Trial product 8 — Buffering agent: Disodium hydrogen phosphate dihydrate 5.34 mg/mL Isotonic agent: NaCl 6.72 mg/mL
Other: Trial product 9 — Buffering agent: Tris 2.4 mg/mL Isotonic agent: Propylene glycol 19 mg/mL
Other: Trial product 10 — Buffering agent: Glutamic acid 0.74 mg/mL Isotonic agent: Glycerol 24.0 mg/mL
Other: Trial product 10 — Buffering agent: Sodium Acetate, trihydrate 0.68 mg/mL Isotonic agent: Glycerol 24.0 mg/mL
Other: Trial product 12 — Buffering agent: Glutamic acid 0.46 mg/mL, Disodium hydrogen phosphate, dihydrate 2.00 mg/mL Isotonic agent: Glycerol 15 mg/mL, NaCl 2.5 mg/mL

SUMMARY:
The purpose of this study is to investigate different solutions used to inject drugs under the skin. The solutions used in the study do not contain the drugs they will be used for, but they do contain excipients, which are inactive substances added to drug solutions to ensure the stability (shelf life and correct activity) of the drug product. The excipients are considered 'inactive substances' compared to the drug, but they may cause an undesirable effect at the injection site in the form of pain. However, their pain-causing potential has never been tested in a systematic way. The purpose of the study is to determine if there is a difference in the injection site pain experience after an injection under the skin (subcutaneous) with 12 different study products. These study products are excipient solutions, which are substances in medications next to the active substance. None of the 12 products include active medication. This study will be performed in 108 healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 69 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) equal to or above 25.0 and below 30.0 kg/m^2.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG), and clinical laboratory tests performed during the screening visit, as judged by the Investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant within 1 week of Day 2 or is of childbearing potential and not using highly effective contraceptive methods.
* Any disorder which in the Investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Glycated haemoglobin (HbA1c) equal to or above 6.5 % (48 mmol/mol) at screening.
* Use of prescription medicinal products or non-prescription drugs or herbal products, except routine vitamins, topical medication (when not used in the abdominal area), contraceptives or occasional use of paracetamol (not allowed within 24 hours prior to Trial Product administration), within 14 days prior to Day 1.
* Average intake of more than 21 units of alcohol per week for male subjects and more than 14 units per week for female subjects: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits.
* Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening and admission to the clinical research centre.
* Use of tobacco and nicotine products, defined as any of the below:
* Smoking more than 1 cigarette or the equivalent per day on average.
* Not able or willing to refrain from smoking and use of nicotine substitute products during the in-house period.
* Subject is not able to understand and read English or Dutch, or subject is not able to understand and comply with the trial requirements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Intensity of injection site pain | 1 min after each injection (Day 1 and Day 2)
  mm on a 100 mm horizontal visual-analogue scale (where 0 mm
  = no pain, 100 mm = unbearable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosur (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com